CLINICAL TRIAL: NCT02078219
Title: A Randomized, Double-Blind, Multicenter, Placebo-Controlled, Parallel Group, 24-Week Phase II Study to Evaluate Efficacy and Safety of RDEA3170 5 mg, 7.5 mg, 10 mg, 12.5 mg and 15 mg Versus Placebo and Open-Label Allopurinol 200 mg as a Reference Arm in Japanese Patients With Gout or Asymptomatic Hyperuricemia
Brief Title: Phase II Dose Finding Study of RDEA3170 Versus Placebo in Japanese Patients With Gout or Asymptomatic Hyperuricemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5491C00001; RDEA3170-203 (Other: Ardea Biosciences, Inc.)
Record Dates: First submitted 2014-02-26; First posted 2014-03-05 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-08

CONDITIONS: Gout and Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — verinurad; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- RDEA3170 1 (Experimental): RDEA3170 5mg followed by RDEA3170 7.5mg
  Interventions: Drug: RDEA3170
- RDEA3170 2 (Experimental): RDEA3170 10mg followed by RDEA3170 12.5mg
  Interventions: Drug: RDEA3170
- RDEA3170 3 (Experimental): RDEA3170 12.5mg followed by RDEA3170 15mg
  Interventions: Drug: RDEA3170
- RDEA3170 4 (Placebo Comparator): RDEA3170 Placebo
  Interventions: Drug: Placebo
- Allopurinol (Other): Allopurinol 200mg
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: RDEA3170 — Oral Treatment
  Arms: RDEA3170 1; RDEA3170 2; RDEA3170 3
Drug: Allopurinol — Oral Treatment
  Other Names: Allopurinol 200mg Sawai
  Arms: Allopurinol
Drug: Placebo — Oral Treatment
  Arms: RDEA3170 4

SUMMARY:
This study is to examine the hypothesis that administration of RDEA3170 to Japanese patients with gout or asymptomatic hyperuricemia in doses of 5 mg, 7.5 mg, 10 mg, 12.5 mg and 15 mg once daily, respectively will result in greater reduction of sUA compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets any of the following criteria and with sUA ≤10.0 mg/dL:

  1. sUA level of >7.0 mg/dL at 7 days prior to baseline with gout;
  2. sUA level of ≥8.0 mg/dL at 7 days prior to baseline without gout but with complications (hypertension, ischemic heart disease, diabetes, metabolic syndrome);
  3. sUA level of ≥9.0 mg/dL at 7 days prior to baseline without gout and complications.

Exclusion Criteria:

* Subject with an acute gout flare that has not resolved at least 14 days prior to the baseline visit.
* Subject has a history or suspicion of kidney stones.
* Subject has an estimated creatinine clearance <60 mL/min calculated by the Cockcroft Gault formula
* Subject is receiving strong or moderate CYP3A inhibitors

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-01-05 (Actual); Primary Completion 2015-03-13 (Actual); Study Completion 2015-03-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Japan (9):
  - Research Site, Chofu-shi
  - Research Site, Fukuoka
  - Research Site, Kitakyushu-shi
  - Research Site, Matsudo-shi
  - Research Site, Noda
  - Research Site, Ōta-ku
  - Research Site, Saitama-shi
  - Research Site, Sendai
  - Research Site, Shinagawa-ku

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 381 subjects who were screened in the study, 204 were randomized into one of the treatment groups. All 204 randomized subjects received at least 1 dose of randomized study medication. The first patient was enrolled on 11 March 2014 and the last enrolled patient completed the Last visit on 13 March 2015.
Pre-assignment Details: 204 were randomized into one of the following treatment groups; allopurinol, placebo, RDEA3170 Group 1, Group 2 and Group 3. Of the enrolled subjects, 177 were withdrawn prior to randomization because of 'eligibility criteria not fulfill' (176 subjects) or 'patient decision' (1 subject).
Groups:
- Allopurinol 200 mg Treatment Group: 100 mg qd for 4 weeks and allopurinol 100 mg bid for 20 weeks
- RDEA3170 Placebo Treatment Group: RDEA3170 matching placebo qd for 24 weeks
- RDEA3170 Treatment Group 1: RDEA3170 2.5 mg once daily (qd) for 4 weeks followed by RDEA3170 5 mg qd for 12 weeks followed by RDEA3170 7.5 mg qd for 8 weeks
- RDEA3170 Treatment Group 2: RDEA3170 2.5 mg qd for 4 weeks followed by RDEA3170 5 mg qd for 4 weeks followed by RDEA3170 10 mg qd for 8 weeks followed by RDEA3170 12.5 mg qd for 8 weeks
- RDEA3170 Treatment Group 3: RDEA3170 2.5 mg qd for 4 weeks followed by RDEA3170 5 mg qd for 4 weeks followed by RDEA3170 12.5 mg qd for 8 weeks followed by RDEA3170 15 mg qd for 8 weeks
Period: Overall Study
Arm/Group | Allopurinol 200 mg Treatment Group | RDEA3170 Placebo Treatment Group | RDEA3170 Treatment Group 1 | RDEA3170 Treatment Group 2 | RDEA3170 Treatment Group 3
Started | 41 | 40 | 41 | 41 | 41
Completed | 38 | 36 | 35 | 37 | 39
Not Completed | 3 | 4 | 6 | 4 | 2
Not completed — Other | 2 | 2 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: No subject was excluded from the safety and efficacy analysis sets. Some data points of 3 subjects who have incompliance were excluded from the PK analyses due to incorrect dose of RDEA3170
Groups:
- Total: Total of all reporting groups
Arm/Group | Allopurinol 200 mg Treatment Group | RDEA3170 Placebo Treatment Group | RDEA3170 Treatment Group 1 | RDEA3170 Treatment Group 2 | RDEA3170 Treatment Group 3 | Total
Number analyzed (Participants) | 41 | 40 | 41 | 41 | 41 | 204
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.0 (10.6) | 54.5 (10.3) | 51.3 (9.3) | 52.7 (10.0) | 52.3 (10.7) | 52.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1 | 2 | 4
  Male | 41 | 39 | 41 | 40 | 39 | 200

OUTCOME MEASURES:

1. Primary Outcome: Percent Changes of Serum Uric Acid Levels From Baseline Levels
Description: The primary objective of the study is to compare percent changes of serum uric acid levels from baseline levels after 16 weeks of dosing between RDEA3170 treatment groups and the placebo treatment group.
Time Frame: Baseline and Week 16
Population: Efficacy analysis set
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Allopurinol 200 mg Treatment Group: Allopurinol 100 mg qd for 4 weeks followed by allopurinol 100 mg twice daily (bid) for 20 weeks
Arm/Group | RDEA3170 Treatment Group 1 | RDEA3170 Treatment Group 2 | RDEA3170 Treatment Group 3 | RDEA3170 Placebo Treatment Group | Allopurinol 200 mg Treatment Group
Number analyzed (Participants) | 41 | 41 | 41 | 40 | 41
Percent change | -30.93 (17.80) | -49.91 (18.38) | -54.32 (13.40) | -2.05 (9.29) | -39.09 (11.54)
Statistical Analysis 1: Comparison: RDEA3170 Treatment Group 1 vs RDEA3170 Placebo Treatment Group; Test type: Superiority or Other; p < 0.0001, ANCOVA, LOCF; Mean Difference (Final Values) = -29.28, 95% CI 2-sided [-36.99 to -21.57]
Statistical Analysis 2: Comparison: RDEA3170 Treatment Group 2 vs RDEA3170 Placebo Treatment Group; Test type: Superiority or Other; p < 0.0001, ANCOVA, LOCF; Mean Difference (Final Values) = -49.25, 95% CI 2-sided [-56.97 to -41.52]
Statistical Analysis 3: Comparison: RDEA3170 Treatment Group 3 vs RDEA3170 Placebo Treatment Group; Test type: Superiority or Other; p < 0.0001, ANCOVA, LOCF; Mean Difference (Final Values) = -53.33, 95% CI 2-sided [-61.00 to -45.67]

2. Secondary Outcome: Percentage of Subjects With a Serum Uric Acid Level ≤6.0 mg/dL
Description: To compare the percentage of subjects whose serum uric acid levels are ≤ 6.0 mg/dL between RDEA3170 treatment groups and the placebo treatment group at each study visit
Time Frame: Weeks 1,2,4,6,8,10,12,16,18,20,24
Population: Efficacy analysis set
Measure: Number; unit: % subjects
Arm/Group | RDEA3170 Treatment Group 1 | RDEA3170 Treatment Group 2 | RDEA3170 Treatment Group 3 | RDEA3170 Placebo Treatment Group | Allopurinol 200 mg Treatment Group
Number analyzed (Participants) | 41 | 41 | 41 | 40 | 41
% subjects
  Week 1 | 26.8 | 31.7 | 39.0 | 0 | 19.5
  Week 2 | 29.3 | 34.1 | 34.1 | 0 | 19.5
  Week 4 | 26.8 | 31.7 | 39.0 | 0 | 17.1
  Week 6 | 70.7 | 61.0 | 82.9 | 0 | 73.2
  Week 8 | 53.7 | 56.1 | 78.0 | 0 | 65.9
  Week 10 | 46.3 | 78.0 | 92.7 | 0 | 61.0
  Week 12 | 53.7 | 85.4 | 92.7 | 0 | 75.6
  Week 16 | 51.2 | 95.1 | 97.6 | 0 | 78.0
  Week 18 | 63.4 | 92.7 | 95.1 | 0 | 73.2
  Week 20 | 61.0 | 82.9 | 92.7 | 0 | 78.0
  Week 24 | 68.3 | 82.9 | 87.8 | 0 | 75.6

3. Secondary Outcome: Percent Change in sUA
Description: To compare percent change in sUA at each study visit.
Time Frame: Baseline, Weeks 1,2,4,6,8,10,12,16,18,20,24
Population: Efficacy analysis set
Measure: Mean (Standard Deviation); unit: % Change
Arm/Group | RDEA3170 Treatment Group 1 | RDEA3170 Treatment Group 2 | RDEA3170 Treatment Group 3 | RDEA3170 Placebo Treatment Group | Allopurinol 200 mg Treatment Group
Number analyzed (Participants) | 41 | 41 | 41 | 40 | 41
% Change
  Week 1 | -19.72 (10.93) | -20.29 (17.51) | -19.93 (22.98) | -0.25 (8.57) | -20.74 (7.72)
  Week 2 | -21.03 (11.87) | -20.28 (16.87) | -20.93 (10.68) | -0.53 (7.20) | -20.80 (9.37)
  Week 4 | -22.95 (10.86) | -19.66 (17.24) | -24.21 (10.69) | 0.97 (8.70) | -20.60 (8.83)
  Week 6 | -32.05 (13.05) | -31.26 (19.83) | -35.24 (10.74) | -0.01 (9.86) | -37.06 (8.72)
  Week 8 | -27.94 (16.54) | -30.19 (19.22) | -32.11 (13.96) | 0.55 (9.50) | -36.51 (11.14)
  Week 10 | -24.69 (18.81) | -37.61 (18.35) | -44.38 (12.33) | -0.27 (9.53) | -33.42 (11.28)
  Week 12 | -28.08 (18.22) | -45.77 (17.94) | -51.17 (16.19) | 0.43 (7.89) | -37.96 (10.65)
  Week 16 | -30.93 (17.80) | -49.91 (18.38) | -54.32 (13.40) | -2.05 (9.29) | -39.09 (11.54)
  Week 18 | -32.94 (18.11) | -49.04 (19.19) | -54.70 (13.32) | -2.86 (8.55) | -38.59 (10.32)
  Week 20 | -32.96 (18.69) | -47.20 (21.46) | -53.60 (12.92) | -2.27 (8.76) | -38.00 (11.11)
  Week 24 | -35.73 (19.49) | -47.34 (21.39) | -54.46 (18.97) | -4.67 (10.36) | -37.77 (11.47)

4. Secondary Outcome: Absolute Change of Serum Uric Acid Levels From Baseline Levels
Description: To compare the absolute change of serum uric acid levels from baseline levels
Time Frame: Baseline, Weeks 1,2,4,6,8,10,12,16,18,20,24
Population: Efficacy analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | RDEA3170 Treatment Group 1 | RDEA3170 Treatment Group 2 | RDEA3170 Treatment Group 3 | RDEA3170 Placebo Treatment Group | Allopurinol 200 mg Treatment Group
Number analyzed (Participants) | 41 | 41 | 41 | 40 | 41
mg/dL
  Week 1: number analyzed (Participants) | 41 | 41 | 41 | 40 | 40
  Week 1 | -1.68 (1.01) | -1.74 (1.48) | -1.68 (2.10) | -0.05 (0.77) | -1.82 (0.73)
  Week 2 | -1.81 (1.11) | -1.75 (1.45) | -1.78 (0.98) | -0.07 (0.64) | -1.83 (0.90)
  Week 4 | -2.01 (1.09) | -1.72 (1.48) | -2.07 (1.01) | 0.06 (0.76) | -1.83 (0.89)
  Week 6 | -2.78 (1.34) | -2.66 (1.73) | -3.00 (1.09) | -0.04 (0.81) | -3.26 (0.93)
  Week 8 | -2.44 (1.48) | -2.61 (1.75) | -2.74 (1.23) | 0.02 (0.85) | -3.22 (1.09)
  Week 10 | -2.19 (1.65) | -3.22 (1.78) | -3.75 (1.19) | -0.06 (0.79) | -2.96 (1.13)
  Week 12 | -2.44 (1.56) | -3.85 (1.62) | -4.33 (1.45) | 0.02 (0.70) | -3.35 (1.09)
  Week 16 | -2.67 (1.48) | -4.24 (1.82) | -4.57 (1.28) | -0.22 (0.81) | -3.44 (1.10)
  Week 18 | -2.86 (1.54) | -4.17 (1.82) | -4.62 (1.27) | -0.27 (0.75) | -3.40 (1.06)
  Week 20 | -2.87 (1.61) | -3.98 (1.97) | -4.52 (1.15) | -0.22 (0.75) | -3.35 (1.15)
  Week 24 | -3.10 (1.67) | -3.99 (1.96) | -4.57 (1.64) | -0.42 (0.90) | -3.31 (1.10)

ADVERSE EVENTS:
Time Frame: Adverse Events and serious adverse events will be collected from the time of informed consent throughout the treatment period and the follow-up period.
Arm/Group | Allopurinol 200 mg Treatment Group | RDEA3170 Placebo Treatment Group | RDEA3170 Treatment Group 1 | RDEA3170 Treatment Group 2 | RDEA3170 Treatment Group 3
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/40 | 1/41 | 1/41 | 0/41
Other Adverse Events (participants affected / at risk) | 22/41 | 23/40 | 26/41 | 26/41 | 21/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Allopurinol 200 mg Treatment Group (N=41) | RDEA3170 Placebo Treatment Group (N=40) | RDEA3170 Treatment Group 1 (N=41) | RDEA3170 Treatment Group 2 (N=41) | RDEA3170 Treatment Group 3 (N=41)
Silent myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Allopurinol 200 mg Treatment Group (N=41) | RDEA3170 Placebo Treatment Group (N=40) | RDEA3170 Treatment Group 1 (N=41) | RDEA3170 Treatment Group 2 (N=41) | RDEA3170 Treatment Group 3 (N=41)
Nasopharyngitis (Infections and infestations) | 7 | 7 | 9 | 8 | 6
Pharyngitis (Infections and infestations) | 2 | 0 | 2 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 1
Chronic pigmented purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 2
Hypertension (Vascular disorders) | 2 | 1 | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Contact stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasal vestibulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Dermatitis infected (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Muscle contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Venomous sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Silent myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No